CLINICAL TRIAL: NCT03767036
Title: Single Site Pharmacokinetic Non-interaction Study With Open-label, Randomized, Single-dose, Three-period, Six-sequence, Crossover Design to Compare Tramadol Hydrochloride 25 mg Capsules (Tradol [Trade Mark], Product of Grünenthal Mexico S.A. de C.V.) and Ketorolac Tromethamine 10 mg Tablets (Dolac [Trade Mark], Product of Siegfried Rhein, S.A. de C.V.) Administered Separately and Simultaneously in Healthy Volunteers Under Fasting Conditions
Brief Title: Administration of Tramadol and Ketorolac Separately and Simultaneously to Assess a Potential Pharmacokinetic Interaction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Grünenthal Colombiana S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP8002-01; TRMKTR-01-GRU (Other: Grünenthal); 16-CI-16 053 026 (Registry Identifier: COFEPRIS)
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Pharmacokinetics
Keywords: tramadol; ketorolac; interaction
MeSH Terms: interventions — Tramadol; Ketorolac Tromethamine; Tablets

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, crossover design with three treatment periods and six sequences (A3-A1-A2, A1-A2-A3, A2-A3-A1, A3-A2-A1, A1-A3-A2, A2-A1-A3) with single administration of tramadol (A1), ketorolac (A2) or tramadol and ketorolac (A3). Treatment periods were separated by a washout period of at least 4 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tramadol (Active Comparator): Each participant received an oral dose of tramadol hydrochloride 25 mg (A1, one capsule) under fasting conditions with 250 milliliters (mL) of water.
  Interventions: Drug: Tramadol hydrochloride 25 mg capsule
- Ketorolac (Active Comparator): Each participant received an oral dose of ketorolac 10 mg (A2, one tablet) under fasting conditions with 250 mL of water.
  Interventions: Drug: Ketorolac Tromethamine 10 mg tablet
- Tramadol and ketorolac (Experimental): Each participant received an oral dose of tramadol hydrochloride 25 mg and ketorolac 10 mg simultaneously (A3 = one capsule of A1 + one tablet of A2, test medication) under fasting conditions with 250 mL of water.
  Interventions: Drug: Tramadol hydrochloride 25 mg capsule; Drug: Ketorolac Tromethamine 10 mg tablet

INTERVENTIONS:
Drug: Tramadol hydrochloride 25 mg capsule — Capsule with tramadol hydrochloride 25 mg; Product of Grünenthal de Mexico S.A. de C.V.
  Other Names: Tradol (trade mark)
  Arms: Tramadol; Tramadol and ketorolac
Drug: Ketorolac Tromethamine 10 mg tablet — Tablet with ketorolac tromethamine 10 mg; Product of Siegfried Rhein, S.A. de C.V., Mexico
  Other Names: Dolac (trade mark)
  Arms: Ketorolac; Tramadol and ketorolac

SUMMARY:
Tramadol (Tradol) and ketorolac (Dolac) are marketed products to treat acute pain. This study was performed to determine if both medications can be given to a patient simultaneously without a change of the products' bioavailability.

DETAILED DESCRIPTION:
The primary objective of the study was to compare the bioavailability of tramadol 25 mg and ketorolac 10 mg after oral single-dose administration of the individual components, either separately or simultaneously, in healthy volunteers under fasting conditions, to demonstrate the absence of a pharmacokinetic interaction.

The secondary objective of the study was to evaluate the safety of both drugs when administered separately and simultaneously based on adverse events reported after treatment.

Participants were admitted to the study site for approximately 42 hours (12 hours before and 30 hours after dosing) for each of the 3 treatment periods. A final examination was performed 2 days after completion of the last treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the study will be voluntary and according to the guidelines proposed by the Health General Law (from Mexico), and informed consent will be obtained according to the previously mentioned law. In addition, the study will be conducted according to the ethical principles that have their origin in the Declaration of Helsinki, the current Brazilian regulations, and Good Clinical Practice.
* Only healthy volunteers, men and women aged between 18 and 55 years will be included.
* The body mass index must be between 18.0 and 27.0 kilograms per square meter according to the Quetelet index.
* Women of childbearing potential must be willing to use contraceptive methods (including barrier methods, non-hormonal intra-uterine device, or have a preexistent bilateral tubal ligation) or practice abstinence as a form of lifestyle during the conduct of the study.
* Participants must be healthy as determined by the results of a complete clinical history recorded by the clinical investigational site physicians and the results of the laboratory and other complementary diagnostic tests done by a certified clinical laboratory.
* The allowed limits of variation within normal in the screening visit will be: systolic blood pressure (sitting) 90 to 130 millimeters mercury (mmHg), diastolic blood pressure 60 to 89 mmHg, heart rate between 50 and 100 beats per minute and respiratory rate between 12 and 20 breaths per minute according to the current standard operating procedure. Vital signs will be measured after 5 minutes of resting in a sitting position.
* Laboratory and other examinations to be conducted for the inclusion of participants will be:

  1. Complete blood count: leukocytes, erythrocytes, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, erythrocyte distribution width, platelets, neutrophils, lymphocytes, monocytes, eosinophils, basophils.
  2. Blood chemistry 27 elements: glucose, urea, blood urea nitrogen (BUN), creatinine, BUN/creatinine ratio, uric acid, cholesterol, high-density lipoprotein (HDL) cholesterol, triglycerides, low-density lipoprotein (LDL) cholesterol, non-HDL cholesterol, atherogenic index, total protein, albumin, globulins, albumin/globulin ratio, total bilirubin, direct bilirubin, indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, total alkaline phosphatase, gamma-glutamyl transferase, lactate dehydrogenase, iron, calcium, sodium, potassium, and chloride.
  3. Urinalysis: Physical examination (color, appearance, density); chemical examination (pH, leukocytes, nitrite, protein, glucose, ketones, bilirubin, urobilinogen, hemoglobin); microscopic examination (leukocytes, erythrocytes, dysmorphic erythrocytes, casts, crystals, squamous epithelial cells, tubular renal cells, mucus, bacteria and yeasts).
  4. Hepatitis B screening (Antibody to hepatitis B core antigen [Anti-HBc], antibody to hepatitis B surface antigen [HBs-Ab], antibody to hepatitis B surface antigen [Anti-HBs]) and hepatitis C antibodies.
  5. Human immunodeficiency virus (HIV) test: Antibodies to the human immunodeficiency virus (Anti-HIV 1 and 2).
  6. Venereal disease research laboratory (VDRL) test.
  7. Urine drugs of abuse test at the screening visit and at on Day 0 (day prior to the administration of the IMP.
  8. Alcohol breath test at the screening visit and at on Day 0 (day prior to the administration of the IMP.
  9. Serum pregnancy test (beta-human chorion gonadotropin [ß-HCG]) at the screening visit and the final evaluation as well as a urine pregnancy test (qualitative) at approximately 12 hours prior to the administration of the IMP.
  10. 12-lead electrocardiogram (with a validity not older than 3 months).

Exclusion Criteria:

* Participants with a history of the following diseases: cardiovascular (congestive heart failure, ischemic heart disease, peripheral arterial disease, high blood pressure), neurologic (epilepsy, non-controlled seizures, cerebrovascular disease), renal (creatinine clearance below 30 milliliters per minute), hepatic (severe hepatic failure, active hepatic disease or transaminase increase that exceeds three times the upper limit of normal), pulmonary, muscular, metabolic (dehydration, hypovolemia, hyperlipidemia, diabetes mellitus), gastrointestinal (intestinal inflammatory disease) including constipation, endocrine, hematopoietic or any type of anemia, mental disease, or other organic abnormalities as well as those participants who have had muscular trauma within 21 days previous to the study will also be excluded.
* Participants who require any kind of medication during the course of the study, apart from the IMP.
* Participants with a history of dyspepsia, gastritis, esophagitis, duodenal or gastric ulcer, active or recurring gastrointestinal perforation or hemorrhage.
* Current or recent (within 14 days prior to administration of the study medication) use of monoamine oxidase inhibitors (MAOIs).
* Current use of acetylsalicylic, other non-steroidal anti-inflammatory drugs (NSAIDs), pentoxifylline and probenecid.
* Participants with a history of hypersensibility to aspirin and other NSAIDs.
* History of major surgeries (cranial surgery, thorax, abdomen or extensive surgeries in extremity requiring the use of general or regional anesthesia and/or respiratory support) within 3 months prior to the study.
* Participants with a history of asthma, acute rhinitis, nasal polyps, angioneurotic edema, urticarial and allergy-type reactions associated with NSAIDs.
* Participants who have been exposed to medications known to be hepatic enzyme inducers or inhibitors within 30 days (or 7 half-lives) prior to the start of the study.
* Participants who have taken any type of medication including vitamin supplements (with or without prescription) or herbal remedies within 30 days (or 7 half-lives) prior to the start of the study.
* Estimated creatinine clearance (CLcr) equal to or below 80 milliliters per minute based on the Cockcroft-Gault formula (for female participants, the result should be multiplied by 0.85): CLcr = (140-age[year])(corporal weight[kg] divided by (72)(creatinine in serum[milligrams per deciliter]). A participant with a creatinine clearance estimated to be 10 percent or less than 80 milliliters per minute can be randomized at the principal investigator's discretion.
* Participants who have been hospitalized for any reason within 6 months prior to the start of the study.
* Participants who have taken IMPs from other investigations within 180 days (6 months) prior to study start.
* Participants with an allergy to the study medication (tramadol or other opioids/ketorolac), any other medication, food, or substance.
* Participants who have consumed alcohol, carbonated beverages and/or beverages that contain methylxanthines (coffee, tea, cocoa, chocolate, mate, cola, etc.), grapefruit juice, or charbroiled foods within 12 hours prior to the start of the hospitalization period as well as participants who have smoked tobacco within 12 hours prior to the study start.
* Participants who have donated or lost more than 450 milliliters (mL) of blood within 60 days prior to study begin.
* Participants with a history of dependence/abuse of alcohol, psychoactive substances within the 2 previous years.
* Participants requiring a special diet for any reason, e.g., vegetarian.
* Participants unable to understand the nature, objectives, and possible consequences of the study.
* Evidence of the participant's uncooperativeness (lack of adherence to the instructions and requirements of the study personnel) during the process of selection for the study.
* Participants with positive test results for drugs of abuse, pregnancy and/or alcohol.
* Participants currently lactating.
* Participants receiving hormonal therapy via any route of administration.
* Participants who are not registered in the Comisión Federal para la Protección contra Riesgos Sanitarios (COFEPRIS) webpage.
* Relationship of subordination between the participants and the investigators.
* Sponsor or clinical research institute employees.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Tramadol: area under the plasma concentration-time curve from 0 to time t (AUC0-t) | Before IMP administration and up to 30 hours thereafter (20 time points in total)
  One blood sample was taken before administration of the investigational medicinal product (IMP) and one sample at each of the following time points: 0.167, 0.25, 0.333, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 5.0, 7.0, 9.0, 12.0, 18.0, 24.0 and 30.0 hours in each period. The quantification of tramadol was done using a validated reversed phase high-performance liquid chromatography-tandem mass spectrometry bioanalytical assay. The AUC0-t was calculated based on plasma concentration-time data (using the actual blood sampling times).
O-desmethyltramadol: area under the plasma concentration-time curve from 0 to time t (AUC0-t) | Before IMP administration and up to 30 hours thereafter (20 time points in total)
  One blood sample was taken before administration of the IMP and one sample at each of the following time points: 0.167, 0.25, 0.333, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 5.0, 7.0, 9.0, 12.0, 18.0, 24.0 and 30.0 hours in each period. The quantification of O-desmethyltramadol was done using a validated reversed phase high-performance liquid chromatography-tandem mass spectrometry bioanalytical assay. The AUC0-t was calculated based on plasma concentration-time data (using the actual blood sampling times).
Ketorolac: area under the plasma concentration-time curve from 0 to time t (AUC0-t) | Before IMP administration and up to 30 hours thereafter (20 time points in total)
  One blood sample was taken before administration of the IMP and one sample at each of the following time points: 0.167, 0.25, 0.333, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 5.0, 7.0, 9.0, 12.0, 18.0, 24.0 and 30.0 hours in each period. The quantification of ketorolac was done using a validated reversed phase high-performance liquid chromatography-tandem mass spectrometry bioanalytical assay. The AUC0-t was calculated based on plasma concentration-time data (using the actual blood sampling times).
Tramadol: maximum plasma concentration (Cmax) | Before IMP administration and up to 30 hours thereafter (20 time points in total)
  One blood sample was taken before administration of the IMP and one sample at each of the following time points: 0.167, 0.25, 0.333, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 5.0, 7.0, 9.0, 12.0, 18.0, 24.0 and 30.0 hours in each period. The quantification of tramadol was done using a validated reversed phase high-performance liquid chromatography-tandem mass spectrometry bioanalytical assay. Cmax was calculated based on plasma concentration-time data (using actual blood sampling times).
O-desmethyltramadol: maximum plasma concentration (Cmax) | Before IMP administration and up to 30 hours thereafter (20 time points in total)
  One blood sample was taken before administration of the IMP and one sample at each of the following time points: 0.167, 0.25, 0.333, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 5.0, 7.0, 9.0, 12.0, 18.0, 24.0 and 30.0 hours in each period. The quantification of O-desmethyltramadol was done using a validated reversed phase high-performance liquid chromatography-tandem mass spectrometry bioanalytical assay. Cmax was calculated based on plasma concentration-time data (using actual blood sampling times).
Ketorolac: maximum plasma concentration (Cmax) | Before IMP administration and up to 30 hours thereafter (20 time points in total)
  One blood sample was taken before administration of the IMP and one sample at each of the following time points: 0.167, 0.25, 0.333, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 5.0, 7.0, 9.0, 12.0, 18.0, 24.0 and 30.0 hours in each period. The quantification of ketorolac was done using a validated reversed phase high-performance liquid chromatography-tandem mass spectrometry bioanalytical assay. Cmax was calculated based on plasma concentration-time data (using actual blood sampling times).

SECONDARY OUTCOMES:
Tramadol: time to maximum plasma concentration (tmax) | Before IMP administration and up to 30 hours thereafter (20 time points in total)
  One blood sample was taken before administration of the IMP and one sample at each of the following time points: 0.167, 0.25, 0.333, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 5.0, 7.0, 9.0, 12.0, 18.0, 24.0 and 30.0 hours in each period. The quantification of tramadol was done using a validated reversed phase high-performance liquid chromatography-tandem mass spectrometry bioanalytical assay. The time to maximum tramadol plasma concentration was calculated based on plasma concentration-time data (using actual blood sampling times).
O-desmethyltramadol: time to maximum plasma concentration (tmax) | Before IMP administration and up to 30 hours thereafter (20 time points in total)
  One blood sample was taken before administration of the IMP and one sample at each of the following time points: 0.167, 0.25, 0.333, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 5.0, 7.0, 9.0, 12.0, 18.0, 24.0 and 30.0 hours in each period. The quantification of O-desmethyltramadol was done using a validated reversed phase high-performance liquid chromatography-tandem mass spectrometry bioanalytical assay. The time to maximum O-desmethyltramadol plasma concentration was calculated based on plasma concentration-time data (using actual blood sampling times).
Ketorolac: time to maximum plasma concentration (tmax) | Before IMP administration and up to 30 hours thereafter (20 time points in total)
  One blood sample was taken before administration of the IMP and one sample at each of the following time points: 0.167, 0.25, 0.333, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 5.0, 7.0, 9.0, 12.0, 18.0, 24.0 and 30.0 hours in each period. The quantification of ketorolac was done using a validated reversed phase high-performance liquid chromatography-tandem mass spectrometry bioanalytical assay. The time to maximum ketorolac plasma concentration was calculated based on plasma concentration-time data (using actual blood sampling times).

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Investigación Farmacológica y Biofarmacéutica, S.A.P.I de C.V. (IFaB), Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No